CLINICAL TRIAL: NCT00326963
Title: A Multicenter, Open-label Study Evaluating the Safety and Efficacy of a New Protease Inhibitor (Darunavir) With Fuzeon® (Enfuvirtide) Plus Background Antiretroviral Regimen in HIV-1 Infected, Triple-class Treatment-experienced Patients
Brief Title: BLQ Study: A Study of a Protease Inhibitor With Fuzeon (Enfuvirtide) in Treatment-Experienced Patients With HIV-1.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Trimeris (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML19712
Record Dates: First submitted 2006-05-16; First posted 2006-05-17 (Estimated); Results first posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide

ARMS (1):
- Enfuvirtide+PI+ARV's (Experimental): Eligible participants received Fuzeon® (enfuvirtide) 90 milligram (mg) subcutaneously (SC) two times a day (bid) for 24 weeks plus new protease inhibitor (PI) (darunavir/ritonavir) plus other investigator-choice antiretrovirals (ARVs). Participants selected their preferred injection device among the following three options: 27 gauge (G) ½" needle/syringe, 31G 8 millimeter (mm) needle/syringe or Biojector 2000 (B2000) needle-free injection device (NFID).
  Interventions: Drug: Background ARVs; Drug: PI; Drug: enfuvirtide [Fuzeon]

INTERVENTIONS:
Drug: Background ARVs — As prescribed
Drug: PI — As prescribed
Drug: enfuvirtide [Fuzeon] — 90mg sc bid

SUMMARY:
This single arm study will evaluate the efficacy, safety and tolerability of a new investigational protease inhibitor (PI) plus background antiretrovirals plus Fuzeon (90mg sc bid) in HIV-1 infected, triple-class treatment-experienced, Fuzeon-naive adults. The new investigational PI will be administered according to the procedures of the early access program in which the patient is enrolled. The anticipated time on study treatment is 3-12 months, and the target sample size is approximately 120 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* seropositive for HIV-1;
* enrolled in an early access program for a new investigational PI;
* naive to Fuzeon, and the investigational PI;
* treatment-experienced with 3 ARV classes of drug (NRTI, NNRTI and PI).

Exclusion Criteria:

* females who are pregnant or breast-feeding;
* evidence of active, untreated opportunistic infection;
* malignancy requiring chemotherapy or radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2006-03; Primary Completion 2007-04 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (34):
- United States (28):
  - Phoenix, Arizona
  - Bakersfield, California
  - Beverly Hills, California
  - Los Angeles, California
  - San Francisco, California
  - Stanford, California
  - Tarzana, California
  - Norwalk, Connecticut
  - Washington D.C., District of Columbia
  - Fort Lauderdale, Florida
  - Orlando, Florida
  - Port Saint Lucie, Florida
  - Decatur, Georgia
  - Macon, Georgia
  - Baltimore, Maryland
  - St Louis, Missouri
  - Newark, New Jersey
  - Somers Point, New Jersey
  - Albany, New York
  - New York, New York
  - Huntersville, North Carolina
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Annandale, Virginia
  - Hampton, Virginia
- Australia (6):
  - Brisbane
  - Carlton
  - Liverpool
  - Melbourne
  - South Yarra
  - Sydney

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 142 participants were enrolled in this study conducted from 6 March 2006 to 20 April 2007 at 33 centers to be investigated in the United States.
Pre-assignment Details: A total of 142 participants were randomized, of which 140 received the study drug. A total of 2 randomized participants did not receive study drug.
Period: Overall Study
Arm/Group | Enfuvirtide+PI+ARV's
Started | 140
Completed | 107
Not Completed | 33
Not completed — Adverse Event | 2
Not completed — Injection site reaction | 1
Not completed — Death | 1
Not completed — Failure to return | 10
Not completed — Withdrawal by Subject | 10
Not completed — Refused treatment / did not cooperate | 5
Not completed — Violation of selection criteria at entry | 2
Not completed — Other protocol violation | 1
Not completed — Administrative / other | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis was performed on all randomized participants including two participants who does not received study drug.
Groups:
- Enfuvirtide+PI+ARV's: Eligible participants received enfuvirtide 90 mg bid, SC injection for 24 weeks plus new PI (darunavir/ritonavir) plus other investigator-choice ARVs. Participants selected their preferred injection device among the following 3 options: 27G ½" needle/syringe, 31G 8 mm needle/syringe or B2000 NFID.
Arm/Group | Enfuvirtide+PI+ARV's
Number analyzed (Participants) | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (7.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 122

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Human Immunodeficiency Virus Type 1 (HIV-1) Ribonucleic Acid (RNA) Viral Load <50 Copies/mL
Description: Blood samples for HIV-1 RNA viral load measurement were collected at the Week 24 clinic visit. The number of participants with HIV-1 RNA viral load results <50 copies/mL is reported.
Time Frame: Week 24
Population: Analysis was performed on the Intent-to-treat (ITT) Population. The ITT Population included enrolled participants who received at least one dose of study medication and had at least one post baseline efficacy assessment.
Measure: Number; unit: participants
Arm/Group | Enfuvirtide+PI+ARV's
Number analyzed (Participants) | 131
participants
  Imputation by neighboring visit values; At Week 24 | 79
  Without imputation by neighboring visit;At Week 24 | 78

2. Primary Outcome: Percentage of Participants With HIV-1 RNA Viral Load <50 Copies/mL
Description: Blood samples for HIV-1 RNA viral load measurement were collected at the Week 24 clinic visit. The percentage of participants with HIV-1 RNA results <50 copies/mL is reported.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number (97.5% Confidence Interval); unit: Percentage of Participants
Arm/Group | Enfuvirtide+PI+ARV's
Number analyzed (Participants) | 131
Percentage of Participants
  Imputation by neighboring visit values; At Week 24 | 60.3 [51.5 to NA] — We reported lower confidence limit from 1-sided 97.5% confidence interval which was constructed using the normal approximation to the binomial distribution therefore, upper limit is not required. Hence, presented as NA.
  Without imputation by neighboring visit;At Week 24 | 59.5 [50.8 to NA] — We reported lower confidence limit from 1-sided 97.5% confidence interval which was constructed using the normal approximation to the binomial distribution therefore, upper limit is not required. Hence, presented as NA.

3. Secondary Outcome: Number of Participants With HIV-1 RNA Viral Load <50 Copies/mL
Description: Blood samples for HIV-1 RNA viral load measurement were collected at the Week 4 and Week 12 clinic visit. The number of participants with HIV-1 RNA results <50 copies/mL is reported.
Time Frame: Week 4 and 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Enfuvirtide+PI+ARV's
Number analyzed (Participants) | 131
participants
  Imputation by neighboring visit values; At Week 4 | 28
  Without imputation by neighboring visit; At Week 4 | 28
  Imputation by neighboring visit values; At Week 12 | 64
  Without imputation by neighboring visit;At Week 12 | 63

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA Viral Load <50 Copies/mL
Description: Blood samples for HIV-1 RNA viral load measurement were collected at the Week 4 and Week 12 clinic visit. The percentage of participants with HIV-1 RNA Viral Load results <50 copies/mL is reported.
Time Frame: Week 4 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Enfuvirtide+PI+ARV's
Number analyzed (Participants) | 131
Percentage of Participants
  Imputation by neighboring visit values; At Week 4 | 21.4 [14.0 to 28.8]
  Without imputation by neighboring visit; At Week 4 | 21.4 [14.0 to 28.8]
  Imputation by neighboring visit values; At Week 12 | 48.9 [39.9 to 57.8]
  Without imputation by neighboring visit;At Week 12 | 48.1 [39.2 to 57.0]

5. Secondary Outcome: Number of Participants With HIV-1 RNA Viral Load <400 Copies/mL
Description: Blood samples for HIV-1 RNA viral load measurement were collected at the Week 4, Week 12, and Week 24 clinic visit. The number of participants with HIV-1 RNA Viral Load results <400 copies/mL is reported.
Time Frame: Weeks 4, 12, and 24
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Enfuvirtide+PI+ARV's
Number analyzed (Participants) | 131
participants
  Imputation by neighboring visit values; At Week 4 | 74
  Imputation by neighboring visit values; At Week 12 | 89
  Imputation by neighboring visit values; At Week 24 | 95
  Without imputation by neighboring visit;At Week 4 | 74
  Without imputation by neighboring visit;At Week 12 | 88
  Without imputation by neighboring visit;At Week 24 | 94

6. Secondary Outcome: Percentage of Participants With HIV-1 RNA Viral Load <400 Copies/mL
Description: as for outcome 5
Time Frame: Weeks 4, 12, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Enfuvirtide+PI+ARV's
Number analyzed (Participants) | 131
Percentage of participants
  Imputation by neighboring visit values; At Week 4 | 56.5 [47.6 to 65.4]
  Imputation by neighboring visit values; At Week 12 | 67.9 [59.6 to 76.3]
  Imputation by neighboring visit values; At Week 24 | 72.5 [64.5 to 80.5]
  Without imputation by neighboring visit;At Week 4 | 56.5 [47.6 to 65.4]
  Without imputation by neighboring visit;At Week 12 | 67.2 [58.8 to 75.6]
  Without imputation by neighboring visit;At Week 24 | 71.8 [63.7 to 79.8]

7. Secondary Outcome: Change From Baseline in Log 10 Plasma HIV-1 RNA Viral Load
Description: Summary statistics for change from baseline in plasma HIV-1 RNA count were presented. Change from baseline in plasma HIV-1 RNA count was derived as follows: Change from baseline = (plasma HIV-1 RNA count at Week X) - (plasma HIV-1 RNA count at baseline).
Time Frame: Baseline (Day 1), Weeks 4, 12, and 24
Population: Analysis was performed on the Intent-to-treat (ITT) Population. The ITT Population included enrolled participants who received at least one dose of study medication and had at least one post baseline efficacy assessment. Maximum number of participants available at the particular time point were analysed and reported.
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Enfuvirtide+PI+ARV's
Number analyzed (Participants) | 116
copies/mL
  At Week 4; n = 116 | -2.22 (0.783)
  At Week 12; n = 109 | -2.51 (0.961)
  At Week 24; n = 107 | -2.61 (1.099)

8. Secondary Outcome: Number of Participants With Any Adverse Event (AE) and Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAEs are defined as those events that were fatal or immediately life-threatening, and those events that resulted in hospitalization; prolonged an existing hospitalization; resulted in disability; or was a congenital anomaly.
Time Frame: Up to Week 28
Population: Analysis was performed on the Safety Population. The Safety Population included all the participants who received at least one dose of trial medication and had a safety follow-up.
Measure: Number; unit: participants
Arm/Group | Enfuvirtide+PI+ARV's
Number analyzed (Participants) | 137
participants
  Number of participants with at least one AE | 15
  Number of participants with at least one SAE | 13

9. Secondary Outcome: Change From Baseline in CD4+ Lymphocyte Count
Description: Summary statistics for change from baseline in CD4+ lymphocyte count were presented . Change from baseline in CD4+ lymphocyte count was derived as follows: Change from baseline = (CD4+ count at Week X) - (CD4+ count at baseline).
Time Frame: Baseline (Day 1), Weeks 4, 12, and 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Enfuvirtide+PI+ARV's
Number analyzed (Participants) | 114
cells/mm^3
  At Week 4; n = 114 | 56 (93.6)
  At Week 12; n = 109 | 83 (112.9)
  At Week 24; n = 105 | 89 (103.4)

10. Secondary Outcome: Number of Participants Meeting Virologic Failure Criteria
Description: The participant was considered as virologic failure at Week 12 clinic visit if patient achieved HIV-RNA <50 copies/mL at Week 4, and HIV-RNA > 50 copies/mL at Week 12, and HIV-RNA >50 copies/mL confirmed at 2 to 4 weeks after Week 12 or if participants failed to achieve a viral load decrease from baseline greater or equal to 0.5 log10 at Week 12 and failed to achieve a viral load decrease from baseline greater or equal to 0.5 log10 confirmed at 2 to 4 weeks after Week 12. The participant was considered as virologic failure at Week 24 clinic visit if participant achieved HIV-RNA <50 copies/mL at week 12, and HIV-RNA >50 copies/mL at week 24/early discontinuation, and HIV-RNA >50 copies/mL confirmed at 2 to 4 weeks after week 24/early discontinuation or HIV-RNA >50 copies/mL at any time up to week 24 and HIV-RNA >50 copies/mL confirmed at 2 to 4 weeks after week 24/early discontinuation.
Time Frame: Weeks 12 and 24
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Enfuvirtide+PI+ARV's
Number analyzed (Participants) | 131
participants
  Confirmed Failure; At Week 12 | 2
  Confirmed Failure; At Week 24 | 10
  Suspected Failure; At Week 12 | 19
  Suspected Failure; At Week 24 | 45

11. Secondary Outcome: Percentage of Participants Meeting Virologic Failure Criteria
Description: as for outcome 10
Time Frame: Weeks 12 and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Enfuvirtide+PI+ARV's
Number analyzed (Participants) | 131
Percentage of participants
  Confirmed Failure; At Week 12 | 1.5
  Confirmed Failure; At Week 24 | 7.6
  Suspected Failure; At Week 12 | 14.5
  Suspected Failure; At Week 24 | 34.4

12. Secondary Outcome: Number of Participants Adhering to Enfuvirtide (ENF)
Description: Adherence to ENF treatment regimen was calculated using the participant's response to the query on the "Participant Adherence Questionnaire case report form (CRF)" about injections incomplete or missed in the last 4 days preceding the study visit. The percentage adherence to the ENF regimen at each study visit is given by: % Adherence = ([8 - the number of doses missed] / 8) x 100. The number and percentage of participants adhering to the ENF regimen were presented by adherence category (100%, ≥95%, ≥90% and ≥85%) at Weeks 4, 12, and 24.
Time Frame: Weeks 4, 12, and 24
Population: Analysis was performed on the Intent-to-treat (ITT) Population.The ITT Population included enrolled participants who received at least one dose of study medication and had at least one post baseline efficacy assessment. Maximum number of participants available at the particular time point were analysed and reported.
Measure: Number; unit: participants
Arm/Group | Enfuvirtide+PI+ARV's
Number analyzed (Participants) | 125
participants
  100%; At Week 4; n = 125 | 108
  ≥95%; At Week 4; n = 125 | 108
  ≥90%; At Week 4; n = 125 | 108
  ≥85%; At Week 4; n = 125 | 119
  100%; At Week 12; n = 113 | 98
  ≥95%; At Week 12; n = 113 | 98
  ≥90%; At Week 12; n = 113 | 98
  ≥85%; At Week 12; n = 113 | 106
  100%; At Week 24; n = 93 | 79
  ≥95%; At Week 24; n = 93 | 79
  ≥90%; At Week 24; n = 93 | 79
  ≥85%; At Week 24; n = 93 | 87

13. Secondary Outcome: Percentage of Participants Adhering to ENF
Description: as for outcome 12
Time Frame: Weeks 4, 12, and 24
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Enfuvirtide+PI+ARV's
Number analyzed (Participants) | 125
Percentage of Participants
  100%; At Week 4; n = 125 | 86.4
  ≥95%; At Week 4; n = 125 | 86.4
  ≥90%; At Week 4; n = 125 | 86.4
  ≥85%; At Week 4; n = 125 | 95.2
  100%; At Week 12; n = 113 | 86.7
  ≥95%; At Week 12; n = 113 | 86.7
  ≥90%; At Week 12; n = 113 | 86.7
  ≥85%; At Week 12; n = 113 | 93.8
  100%; At Week 24; n = 93 | 84.9
  ≥95%; At Week 24; n = 93 | 84.9
  ≥90%; At Week 24; n = 93 | 84.9
  ≥85%; At Week 24; n = 93 | 93.5

14. Secondary Outcome: Number of Participants With 1 or More Injection Site Reactions Meeting the Criteria of an Serious Adverse Event
Description: Injection site reactions (ISRs) referred to any localized sign or symptom, including erythema, induration, pruritus, nodules, ecchymosis (degree of bruising/ discoloration), and pain/discomfort. Injection site reactions were monitored by trained study personnel at weeks 1, 4, 12, 16, and 24. Interruption of ENF for toxicity management of recurrent local grade 3 or 4 ISRs until the sign or symptom resolved to grade 2 was at the discretion of the investigator. Any individual injection site signs or symptoms meeting the criteria for a serious adverse event (SAE) had to be reported as an SAE. In the event of a serious ISR, the participant was to immediately discontinue ENF and withdraw from the study. If the participant was not already hospitalized, serious ISRs required a clinic visit within 72 hours of the event.
Time Frame: Week 1 to Week 24
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Enfuvirtide+PI+ARV's
Number analyzed (Participants) | 137
participants | 0

15. Secondary Outcome: Percentage of Participants With 1 or More Injection Site Reactions Meeting the Criteria of an Serious Adverse Event
Description: as for outcome 14
Time Frame: Week 1 to Week 24
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Enfuvirtide+PI+ARV's
Number analyzed (Participants) | 137
Percentage of participants | 0

16. Secondary Outcome: Descriptive Summary of ISR Parameters (ie, Severity and Frequency of Pain and Symptoms) by Injection Device Based on an ISR Grading Tool.
Description: Injection site reactions (ISRs) referred to any localized sign or symptom, including erythema, induration, pruritus, nodules, ecchymosis (degree of bruising/ discoloration), and pain/discomfort. Injection site reactions were monitored by trained study personnel at weeks 1, 4, 12, 16, and 24. Grades 0 through 4 are a measure of intensity, not seriousness. Thus, a grade 3 or grade 4 sign or symptom could be severe, but not necessarily serious. Only active, ongoing ISR were counted. The maximum severity grade for pain/discomfort since the last visit at any injection site was recorded whether or not the maximum severity of pain/discomfort was ongoing at the time of clinical evaluation.
Time Frame: Week 24
Population: Analysis was performed on the Safety Population. The Safety Population included all the participants who received at least one dose of trial medication and had a safety follow-up. Maximum number of participants available at the particular time point were analysed and reported.
Measure: Number; unit: participants
Groups:
- Enfuride+PI+ARV's: Eligible participants received enfuvirtide 90 mg bid, SC injection for 24 weeks plus new PI (darunavir/ritonavir) plus other investigator-choice ARVs. Participants selected their preferred injection device among the following 3 options: 27G ½" needle/syringe, 31G 8 mm needle/syringe or B2000 NFID.
Arm/Group | Enfuride+PI+ARV's
Number analyzed (Participants) | 110
participants
  Ongoing Pain/Discomfort, Grade 0; n= 110 | 73
  Ongoing Pain/Discomfort, Grade 1; n= 110 | 24
  Ongoing Pain/Discomfort, Grade 2; n= 110 | 11
  Ongoing Pain/Discomfort, Grade 3; n= 110 | 1
  Erythema, Grade 0; n= 110 | 68
  Erythema, Grade 1; n= 110 | 23
  Erythema, Grade 2; n= 110 | 12
  Erythema, Grade 3; n= 110 | 5
  Erythema, Grade 4; n= 110 | 1
  Erythema, Grade 3 & 4; n= 110 | 6
  Induration, Grade 0; n= 110 | 57
  Induration, Grade 1; n= 110 | 12
  Induration, Grade 2; n= 110 | 19
  Induration, Grade 3; n= 110 | 13
  Induration, Grade 4; n= 110 | 8
  Induration, Grade 3 & 4; n= 110 | 21
  Pruritus, Grade 0; n= 110 | 96
  Pruritus, Grade 1; n= 110 | 13
  Pruritus, Grade 2; n= 110 | 0
  Pruritus, Grade 3; n= 110 | 0
  Nodules and Cysts, Grade 0; n= 110 | 90
  Nodules and Cysts, Grade 1; n= 110 | 8
  Nodules and Cysts, Grade 2; n= 110 | 3
  Nodules and Cysts, Grade 3; n= 110 | 8
  Nodules and Cysts, Grade 4; n= 110 | 0
  Nodules and Cysts, Grade 3 & 4; n= 110 | 8
  Ecchymosis, Grade 0; n= 110 | 82
  Ecchymosis, Grade 1; n= 110 | 13
  Ecchymosis, Grade 2; n= 110 | 6
  Ecchymosis, Grade 3; n= 110 | 6
  Ecchymosis, Grade 4; n= 110 | 2
  Ecchymosis, Grade 3 & 4; n= 110 | 8

17. Secondary Outcome: Number of Participants Discontinuing Study Medication Due to Clinical Adverse Events
Description: The total number and percentage of participants who discontinued the study medication (ENF) due to clinical adverse events (including clinically significant laboratory abnormalities and AIDS Clinical Trials Group (ACTG) grade≥3 laboratory toxicities) were noted and presented.
Time Frame: Up to Week 24
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Enfuvirtide+PI+ARV's
Number analyzed (Participants) | 137
participants
  Total participants with at least one AE | 3
  Upper Gastrointestinal haemorrhage | 1
  Sepsis | 1
  Rash | 1

ADVERSE EVENTS:
Time Frame: Up to Week 28.
Arm/Group | Enfuvirtide+PI+ARV's
Serious Adverse Events (participants affected / at risk) | 13/137
Other Adverse Events (participants affected / at risk) | 0/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enfuvirtide+PI+ARV's (N=137)
Cellulitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Pneumocystis jiroveci Pneumonia (Infections and infestations) | 1
Pneumonia primary atypical (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Renal failure (Renal and urinary disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Upper Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Neutrophil count decreased (Investigations) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Myopathy steroid (Musculoskeletal and connective tissue disorders) | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.